CLINICAL TRIAL: NCT06723600
Title: Effect of Informing Family Members of Patients by Phone Call on Their Anxiety Level During Undergoing Abdominal Cancer Surgery: A Randomized Controlled Trial
Brief Title: Effect of Informing Family Members of Patients During Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Bahar CANDAS ALTINBAS, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Nurse_Anxiety
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Anxiety
Keywords: Anxiety; Informing; Relatives of the Patient; Phone Call; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group relatives of patients will be informed by the nurse during surgery.
  Interventions: Other: Information
- Control Group (No Intervention): The control group will take rutin informing.

INTERVENTIONS:
Other: Information — Nurse-led family member information
  Arms: Experimental Group

SUMMARY:
Psychological and physiological issues encountered by family members due to the intraoperative process are factors that complicate the support and care systems of the patient. It is stated that family members of patients undergoing surgery, especially those who do not have sufficient information about the surgical process, experience stress, anxiety, and concern. The need for nursing interventions aimed at providing information about the surgical process, reducing the anxiety levels of family members during the surgery, and supporting them is emphasized. In this context, the study aims to evaluate the effect of periodically informing family members of patients undergoing abdominal cancer surgery via phone during the surgery on their anxiety levels.

DETAILED DESCRIPTION:
Once the patient scheduled for surgery is taken to the operating room, communication between the family members and the surgical team, as well as the patient, is cut off. Family members who do not have any information about the progress of the surgery experience anxiety during the waiting period. High levels of anxiety can limit the family members' ability to understand and process information, affecting their ability to cope with the situation. The high anxiety experienced by family members during the surgery can reflect onto the patient postoperatively, potentially negatively impacting the patient's adaptation, recovery process, and family relations. It is known that family members of patients undergoing cancer surgery experience a higher level of anxiety. The anxiety emerging during this process leads to various physiological and psychological negative consequences for the family members. It is known that informing family members by nurses during surgery helps reduce their anxiety. In this direction, the primary aim of the study is to determine the effect of periodically informing family members of patients undergoing abdominal cancer surgery via phone during the surgery on their anxiety levels. Additionally, the study will evaluate the satisfaction levels of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Being a first-degree relative who has given consent,
* Being able to understand and speak Turkish,
* Being literate,
* Willing to participate in the study,
* Using a phone,
* Being present in the hospital before, during, and after the surgery.

Exclusion Criteria:

* Having a hearing or speech impairment,
* Having a psychiatric disorder or using psychiatric medication.

Endpoint Criteria:

* Inability to reach the participant when called during the surgery,
* The patient's death during the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Anxiety | During surgery
  The patient's anxiety level 2 hours after the start of the surgical procedure. Self reported anxiety intensity before surgical process that includes on the day of surgery. State-Trait Anxiety Inventory will be used to evaluate the anxiety. The higher the score is the more anxiety.

SECONDARY OUTCOMES:
Satisfaction with Telephone Information Provided During Surgery | Immediately after the surgery.
  The satisfaction levels of family members in the experimental group with the information provided through telephone calls during the surgery will be assessed using the "Evaluation Form for Telephone Information During Surgery," developed by the researcher based on the literature and validated for content.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Candas Altinbas, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Milli Egemenlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No